CLINICAL TRIAL: NCT05895825
Title: A Phase I Study Evaluating the Safety, Tolerability and Pharmacokinetics of EOC237 in Patients With Advanced Solid Tumor
Brief Title: A Study of EOC237 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yiteng Jingang Bio-pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EOC237-X1-101
Record Dates: First submitted 2023-05-12; First posted 2023-06-09 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation (Experimental): In Part 1 (dose escalation) participants with selected advanced solid tumors will receive escalating doses of EOC237 as monotherapy. Participants can receive EOC237 until disease progression, adverse event (AE), or other discontinuation criteria, whichever occurs first.
  Interventions: Drug: EOC237
- Part 2: Food influence-Group 1 (Experimental): Food influence-Group 1: EOC237 was taken orally under fasted conditions, after a 3-day washout period, EOC237 was taken orally under fed conditions.
  Participants can receive EOC237 until disease progression, AE, or other discontinuation criteria, whichever occurs first.
  Interventions: Drug: EOC237
- Part 2: Food influence-Group 2 (Experimental): Food influence-Group 2: EOC237 was taken orally under fed conditions, after a 3-day washout period, EOC237 was taken orally under fasted conditions.
  Participants can receive EOC237 until disease progression, AE, or other discontinuation criteria, whichever occurs first.
  Interventions: Drug: EOC237

INTERVENTIONS:
Drug: EOC237 — EOC237 for orally

SUMMARY:
This research study is studying an investigational drug called EOC237 in Patients With Advanced Solid Tumor.

DETAILED DESCRIPTION:
Part 1 Dose Escalation: an open, single/multiple dose, multi-center phase I study to evaluate the safety, tolerability and pharmacokinetics of EOC237 in Patients With Advanced Solid Tumor.

Part 2 Food influence research: to assess the effect of food on the pharmacokinetics of EOC237, by investigating the bioavailability following single dose administration under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Solid Tumors for which standard curative or palliative measures do not exist or are no longer effective.
* Expected survival≥ 3 months.
* ECOG performance status 0-1.
* Good organ and marrow function.

Exclusion Criteria:

* Patients with a history of severe drug allergic reaction.
* Pregnant or lactating female subjects.
* Uncontrolled, significant intercurrent or recent illness.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per electrocardiogram (ECG)
* Concomitant use of certain medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with dose-limiting toxicity (DLT) | Up to approximately 3 years
  Number of subjects who experienced DLT events during 28 days after first administration of EOC237, divided by the number of DLT evaluable Subjects
Determination of maximum tolerated dose (MTD) | Up to approximately 3 years
the recommended phase 2 dose (RP2D) | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/ Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China